CLINICAL TRIAL: NCT04973579
Title: SIMultaneous Urgent Cardiac Surgery and Endovascular Stroke Prevention Using the Micronet-covered CGUARD Stent in Hemodynamically Compromised Patients at Increased Peri-operative Stroke Risk: SIM-GUARD Study
Brief Title: Simultaneous Cardiac Surgery and Micronet-covered Stent Carotid Revascularization in High Perioperative Stroke Risk Patients
Acronym: SIM-GUARD
Status: Recruiting | Type: Observational
Sponsor: John Paul II Hospital, Krakow (Other)
Responsible Party: Sponsor
Other Study IDs: SIM-GUARD
Record Dates: First submitted 2021-07-13; First posted 2021-07-22 (Actual); Last update posted 2021-07-22 (Actual); Status verified 2021-07

CONDITIONS: Carotid Stenosis; Coronary Artery Disease; Valvular Heart Disease; Myocardial Infarction; Pulmonary Edema With Heart Failure
Keywords: Carotid Stenosis; Coronary Artery Disease, Valvular Disease; Heart Failure, Pulmonary Edema; Single Anesthesia; Simultaneous Procedure
MeSH Terms: conditions — Carotid Stenosis; Coronary Artery Disease; Heart Valve Diseases; Myocardial Infarction; Heart Failure; Pulmonary Edema | interventions — Anesthesia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Simultaneous cardiac surgery and carotid stenting: Patients with Heart Team and NeuroVascular Team recommendation to perform simutaneous (single anaesthesia) carotid artery stenting with MicroNet covered stent (CGuard) including proximal or distal neuroembolic protection and cardiac surgery (CABG or surgical valve replacement / repair procedure)
  Interventions: Procedure: Simutaneous (single anaesthesia) carotid artery stenting with MicroNet covered stent (CGuard) and cardiac surgery (CABG or surgical valve replacement / repair procedure)

INTERVENTIONS:
Procedure: Simutaneous (single anaesthesia) carotid artery stenting with MicroNet covered stent (CGuard) and cardiac surgery (CABG or surgical valve replacement / repair procedure) — The registry enrolls patients qualified for treatment with the methods evaluated in the registry, using routinely applicable procedures and devices.
  In cardiac surgery - surgical treatment systems for advanced ischemic heart disease and/or valvular disease (including - mechanical/biologic heart valves - regulatory approved for routine use and typically used at the Facility.
  In the simultaneous treatment of stroke-threatening carotid artery atherosclerosis - temporary neuroprotection systems (proximal, distal, according to medical indications and local experience) - regulatory approved for routine use and typically used at the center (for over 20 years).
  CGuard anti-embolic mesh stent system - a self-expanding nitinol carotid stent wrapped in MicroNet, which prevents fragments of atherosclerotic plaque from entering the lumen of the carotid artery - approved for routine use and typically used at the Center (over 5 years).

SUMMARY:
Prospective, single-center, clinical registry of patients with symptomatic/critical carotid artery stenosis at risk of stroke coexisting with unstable or multivessel severe coronary artery disease and/or severe valvular heart disease undergoing endovascular treatment of carotid atherosclerosis using a mesh stent in combination with cardiac surgery (coronary artery bypass grafting (CABG) and/or valve surgery). A study involving clinical data evaluation of truly simultaneous treatment outcomes in patients deemed to require carotid revascularization at the time of surgical cardiac intervention (single-stage, simultaneous treatment). An open-label study, without randomization - a single arm study.

Academic Registry - scientific activity of the Faculty of Medicine, Collegium Medicum, Jagiellonian University and John Paul II Hospital.

DETAILED DESCRIPTION:
The coexistence of symptomatic or unstable stroke-threatening carotid atherosclerotic stenosis with cardiac disease requiring urgent / fast-track cardiac surgery (such as advanced unstable or multivessel coronary artery disease, recent myocardial infarction or pulmonary edema, severely impaired myocardial contractility, and/or severe valvular disease requiring surgical treatment) represents a major medical and therapeutic/logistics challenge.

According to current guidelines, in absence of prospective randomized evidence, the most appropriate management strategy for a given patient should be determined by a multispecialty team. In hemodynamically compromised patients sequential treatment (i.e., first carotid stenosis repair followed by surgery or first cardiac surgery followed by carotid stenosis treatment, either surgical or endovascular) is associated with a high risk of cardiac complications in case of first-stage carotid stenosis treatment and a high risk of neurological complications in case of the first-stage cardiac surgery.

In this challenging patient group, we have introduced single-stage, truly simultaneous procedure. The fundament of the strategy is to establish extracorporeal circulation back-up ("CEC standby") prior to the minimally invasive (endovascular) treatment of stroke-threatening carotid artery stenosis in the hybrid room under single anesthesia.

For CAS (proximal or distal protected), in case of suboptimal femoral access (or lack of femoral access), a direct access via carotid artery is used (transcervical or transcarotid revascularization), this is immediately followed by cardiac surgery.

The procedure, each time, follows recommendation of the Multispecialty Team (Heart Team + NeuroVascular Team) as the lowest-deemed risk management in patients with indications for both urgent both carotid revascularization and cardiac surgery. Both carotid and cardiac treatment are performed under single anesthesia with the feasibility of immediate extracorporeal circulation support during carotid revascularization in case of hemodynamic collapse.

Eligibility for treatment is based on the decision (recommendation) of a multidisciplinary Heart Team along with a NeuroVascular Team consisting of a cardiac surgeon, cardiologist, anesthesiologist, angiologist, neurologist, and vascular surgeon, with the concomitant use of routine pharmacotherapy and non-pharmacological prevention - according to current guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Patients eligible for concomitant carotid artery stenting in conjunction with cardiac surgery based on Heart Team and NeuroVascular Team reccomendation and according to local standards of practice.
* Signed informed consent form
* Consent to (routinely performed in this group of patients) follow-up visits and tests performed (routinely) during long-term follow-up
* De novo atherosclerotic lesions or neo-atherosclerosis.
* Symptomatic patients (with a history of ipsilateral transient cerebral ischemia, stroke or amaurosis fugax within the past 6 months) with carotid artery stenosis ≥50% as assessed by NASCET angiography or
* Asymptomatic patients with carotid artery stenosis ≥70-80% as assessed by angiography (NASCET method).
* Coronary angiography-confirmed multivessel disease or left main stem stenosis with the symptoms of unstable angina or non-ST-segment elevation myocardial infarction.
* Severe symptomatic valvular disease detected by echocardiography.

Exclusion Criteria:

* Expected survival time <1 year (e.g., cancer).
* Renal failure with GFR < 20 ml/min/1.73 m2 as calculated by the CKD-EPI formula
* Women who are pregnant (pregnancy test).
* Coagulopathies.
* History of hypersensitivity to a contrast agent that does not respond to pharmacotherapy.
* Total carotid artery occlusion.
* Stent in the carotid artery that protrudes into the aortic arch.
* Anatomic variants that preclude stent implantation.
* Significant stenosis of the common carotid artery proximal to the target lesion.
* Mobile atherosclerotic plaques in the aortic arch.
* Anatomy of the coronary arteries unsuitable for bypass grafting.
* Lack of available vascular material for grafting.
* Porcelain aorta.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All-comers registry of patients with Heart and NeuroVascular Team recommendation for single-stage simultaneous surgical and endovascular procedure.
  The SIM-GUARD single arm registry design and exploratory nature precluded sample size calculation. The number of patients to be enrolled is selected based on the number of procedures at the Center and the average typical size of studies/registries in this field of interventional treatment.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-05-01 (Actual); Primary Completion 2022-05-01 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
Freedom from major clinical complications comprising MACNE (major adverse cardiovascular or neurologic event) at 30 days | 30 days from index procedure
  Freedom from any death, any stroke, and myocardial infarction at 30-day follow-up

SECONDARY OUTCOMES:
Freedom from major clinical complications comprising MACNE at 6 months | At 6 months from index procedure
  Freedom from any death, any stroke, and myocardial infarction at 6 months follow-up
Freedom from major clinical complications comprising MACNE at 12 months | At 12 months from index procedure
  Freedom from any death, any stroke, and myocardial infarction at 12 months follow-up
Procedural success rate for carotid stenting | Periprocedural
  Success of endovascular treatment of carotid artery stenosis i.e. technical success (stent delivery and implantation, withdrawal of stent delivery system, residual stenosis ≤30% of vessel lumen diameter) plus clinical success (procedure without complications).
Technical success | At the procedure completion
  Number of procedures (both carotid and coronary) completed in relation to the number of attempted procedures
Clinical success | Day 2 after procedure
  Number of procedures (both carotid and coronary) completed in relation to the number of attempted procedures in absence of stroke
Rate of arterial access complications | Up to 24 hours post-procedure
  Peri-procedural vascular access complications of carotid artery stenting (pseudoaneurysm of the femoral artery, acute ischemia of the lower limb, massive bleeding from the puncture site) occurring within 24 hours.
Rate of cardiac surgery related complications | Up to 24 hours post-procedure
  Peri-procedural complications associated with cardiac surgery - bleeding requiring re-thoracotomy, cardiac tamponade
Rate of other major peri-procedural complications | Up to 7 days post-procedure
  Other major peri-procedural complications: acute renal failure, systemic infection, respiratory failure requiring prolonged ventilation (>24 hours).
Rate of ipsilateral stroke in the first year | From 31 days till 365 days post-procedure
  Occurence of any ipsilateral stroke
Rate of ipsilateral stroke up to 5 years | From 1 year till 5 years post-procedure
  Occurence of any ipsilateral stroke
Rate of any stroke up to 5 years | Untill 5 years post-procedure
  Occurence of any stroke during registry follow up
Stroke free survival rate up to 1 year | Untill 1 year post-procedure
  Survival without any stroke up to 1 year follow up
Ipsilateral stroke free survival rate up to 1 year | Untill 1 year post-procedure
  Survival without ipsilateral stroke up to 1 year follow up
Stroke free survival rate up to 5 years | Untill 5 year post-procedure
  Survival without any stroke up to 5 year follow up
Ipsilateral stroke free survival rate up to 5 years | Untill 5 year post-procedure
  Survival without ipsilateral stroke up to 5 year follow up
Rate of coronary or carotid restenosis | Untill 5 year post-procedure
  Clinical coronary or carotid restenosis requiring treatment
Rate of cardiac or carotid reintervention | Untill 5 year post-procedure
  Clinically indicated carotid or cardiac reintervention during folow up period
Ultrasound Evaluated Carotid Artery Velocities | After procedure and at 12 months follow up
  Peak Systolic Velocity (PSV) and End Diastolic Velocity (EDV) in the internal carotid/common carotid artery assessed by ultrasound - after the procedure, then at 12 months after the procedure.
Recurrence of angina or valvular heart disease at 30 days and 12 months | At 30 days and 12 months after surgery
  Recurrence of angina or symptomatic valvular heart disease
Recurrence of angina or valvular heart disease up to 5 years | Up to 5 years thereafter after surgery
  Recurrence of angina or symptomatic valvular heart disease
Feasibility of combined treatment | At the procedure completion
  Number of patients actually treated with combined treatment to the number of patients qualified for treatment (excluding deaths in-between)

CONTACTS AND LOCATIONS:
Overall Officials: Piotr Musialek, MD, DPhil, Principal Investigator — Department of Cardiac and Vascular Diseases, John Paul II Hospital
Locations (1):
- Department of Cardiac and Vascular Diseases, John Paul II Hospital, Krakow, Poland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Dzierwa K, Kedziora A, Tekieli L, Mazurek A, Musial R, Dobrowolska E, Stefaniak J, Pieniazek P, Paluszek P, Konstanty-Kalandyk J, Sobczynski R, Kapelak B, Kleczynski P, Brzychczy A, Kwiatkowski T, Trystula M, Piatek J, Musialek P. Endovascular carotid revascularization under open-chest extracorporeal circulation combined with cardiac surgery in unstable patients at increased risk of carotid-related stroke: SIMultaneous urgent cardiac surgery and MicroNet-covered stent carotid revascularization in extreme-risk patients-SIMGUARD Study. J Cardiovasc Surg (Torino). 2023 Dec;64(6):591-607. doi: 10.23736/S0021-9509.23.12896-5. Epub 2023 Dec 11. PMID 38078710